CLINICAL TRIAL: NCT04466761
Title: Phase I Ascending Dose Study of Dietary Supplementation With Glycan Monomers in Healthy Adults
Brief Title: Ascending Glycan Dietary Supplementation in Healthy Adults
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The IRB closed the protocol. PI failed to submit study for continuing review.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1516913
Record Dates: First submitted 2020-06-26; First posted 2020-07-10 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Healthy Individuals
Keywords: Healthy Adults; Dietary supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Cohort 1-4 (Experimental): 60% of subjects per cohort will consume 30-90 grams of dietary supplement daily for 4 weeks, with each successive cohort dosage increasing according to a Fibonacci dose escalation.
  Interventions: Dietary Supplement: Monosaccharide Powder
- Placebo: Cohort 1-4 (Placebo Comparator): 40% of subjects per cohort will consume 30-90 grams of daily placebo for 4 weeks with each successive cohort dosage increasing in parallel to the experimental arm.
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Dietary Supplement: Monosaccharide Powder — Monosaccharide powder dissolved in water.
  Arms: Experimental: Cohort 1-4
Other: Placebo Comparator — Placebo (cellulose powder).
  Arms: Placebo: Cohort 1-4

SUMMARY:
The investigators will conduct a parallel-group, placebo-controlled, randomized, double-blind ascending dose Phase I study of dietary supplementation in healthy individuals to evaluate safety and to determine the pharmacologically effective dose (ED).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-45 years of age
* Patients who are in general good health
* Body Mass Index (BMI) range of 18.5-25
* All individuals must have the ability to provide inform consent

Exclusion Criteria:

* Women who are pregnant, actively nursing, or pregnant within the last year
* Women who are peri-menopausal or post-menopausal
* Women with irregular menstrual cycles (more frequently than every 21 days or lasts longer than 8 days (missed, early, or late periods are also considered signs of an irregular cycle).
* Women on hormonal contraception, including birth control, hormonal intrauterine device, or contraceptive implant
* Past medical history of an autoimmune condition or malignancy, excluding non-melanoma skin cancer
* Individuals with first degree relative with history of an autoimmune condition
* Individuals with cardiovascular, pulmonary, reproductive, endocrine, metabolic, neurologic, gastrointestinal, hematologic, or infectious diseases of any kind
* Individuals with diagnosis of galactosemia or congenital disorders of glycosylation
* Individuals with phenylketonuria
* Individuals currently taking prescription medications, or have taken prescription medications within the last 3 months
* Individuals currently taking over the counter medications
* Individuals currently taking or have taken supplements including herbal, protein or vitamin supplements in the last 3 months (e.g. whey protein, St. John's Wort, green tea supplements, biotin, creatine supplements), excluding multivitamins or essential vitamins
* Individuals with prior history of severe food or drug allergic reactions
* Individuals with a diagnosis of type I or II diabetes mellitus
* Individuals with allergic reaction or adverse reaction to shellfish, N-acetyl glucosamine, galactose, or Spirulina/chlorella/algae supplements
* Individuals with social history of current use of tobacco, alcohol or other drugs
* Individuals with dietary restrictions (vegetarians are permitted to participate in the study) or to whom any of the following dietary habits or characteristics apply (the following exclusion criteria are placed to minimize variability in diet in our study population):

  * Actively dieting or trying to lose weight
  * Vegan diet
  * Consume equal to or greater than 2 cups of tea a day
  * Consume equal to or greater than 4 cups of coffee a day
  * Consume equal to or greater than 3 cups of fruit juice a day
  * Practice intensive exercise patterns (marathon training, workouts >4 hours a day)
  * Consume soda or energy drinks of any amount
  * On a carbohydrate-restricted or "Paleo" diet
  * Calorie-restricted diet (less than 20%-25% of maintenance calories)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-08-06 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Characterize Immunoglobulin fragment crystallization modifications | 4 Weeks
  Use mass spectrometry and RNA sequencing from subject blood samples to characterize site specific glycosylation on Immunoglobulin A, Immunoglobulin M, and Immunoglobulin G.
Identify the maximum effective dose | 16 Weeks
  Identify maximum effective dose of dietary supplement in grams/day.

SECONDARY OUTCOMES:
Assess for potential adverse events | 2 Months after first dose
  Monitor symptoms, severity, and duration of adverse events.
Quantification of enzymatic modifications measured in grams by spectrometry | 6 Months
  The investigators will measure enzymatic changes on glycoproteins in the immune system by spectrometry, i.e., these changes will be measured in grams. Spectometry will allow the investigators to quantify these changes in small detail, and therefore give a better idea of how supplementation can change enzymatic process that then affect the structure, and mass, of glycoproteins.
Flow cytometry to determine the effect of dietary supplementation on the immune system | 6 Months
  Perform flow cytometry on subject blood samples to determine the effect of dietary supplement on immune system. For example, the investigators will note changes to immune cell pro-inflammatory and anti-inflammatory cytokine clusters as translated proteins (measured as height and area of cytokine intensity).
Transcriptome analysis to determine the effect of dietary supplementation on the immune system | 6 Months
  Perform transcriptome analysis on subject blood samples to determine the effect of dietary supplement on immune system. For example, the investigators will note changes to immune cell pro-inflammatory and anti-inflammatory cytokine clusters as RNA (measure on a logarithmic scale per number of reads) to determine the effects of supplementation on both gene transcription and translation.

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No